CLINICAL TRIAL: NCT06093230
Title: An Open-label, Single-dose, Phase I Study to Assess the Pharmacokinetics and Safety of JT001 in Subjects With Mild and Moderate Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Brief Title: A Study in Subjects With Liver Function Injury and Subjects With Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Vinnerna Biosciences Co., Ltd. (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: JT001-007-I
Record Dates: First submitted 2023-09-25; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Subjects With Liver Function Injury; Normal Liver Function Subject
MeSH Terms: interventions — GS-621763

STUDY DESIGN:
Intervention Model Description: Parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): mild liver function impairment group
  Interventions: Drug: Deuremidevir Hydrobromide Tablets
- Group B (Experimental): moderate liver function impairment group
  Interventions: Drug: Deuremidevir Hydrobromide Tablets
- Group C (Experimental): normal liver function subject group
  Interventions: Drug: Deuremidevir Hydrobromide Tablets

INTERVENTIONS:
Drug: Deuremidevir Hydrobromide Tablets — JT001 single dose, 0.3g
  Other Names: JT001

SUMMARY:
Evaluate the pharmacokinetic differences of the main metabolite 116-N1 of JT001 in subjects with mild and moderate liver function impairment and those with normal liver function, providing a basis for formulating clinical medication plans for patients with liver function impairment;

DETAILED DESCRIPTION:
This study adopts a non randomized, open, parallel controlled, single dose experimental design and is divided into three experimental groups: mild liver function impairment group (Group A), moderate liver function impairment group (Group B), and normal liver function subject group (Group C). Subjects in each experimental group took 0.3g of JT001 orally on an empty stomach and collected blood samples before and after administration for pharmacokinetic analysis.

After both groups A and B were enrolled, Group C subjects will be enrolled subsequently and should be matched with subjects with liver function impairment (Group A and Group B) as following:

The average body weight of Group C is within ± 10 kg of the average body weight of the group of subjects with liver function impairment (Groups A and B).

The average age of Group C is within ± 10 years of the average age of the group of subjects with liver function impairment (Groups A and B).

The number of subjects of each gender in Group C is similar to that in the liver function impairment group (A and B groups) (± 1 subject/gender).

The study is divided into three stages: screening period, baseline period, and experimental period.

ELIGIBILITY:
Inclusion Criteria:

1. On the day of signing the informed consent form, the age range is 18 to 70 years (including both ends), both male and female are eligible;
2. Male subjects weighing no less than 50 kg and female subjects weighing no less than 45 kg; Body mass index (BMI) 18-32 kg/m2 (including both ends), where BMI=weight (kg)/height 2 (m2);

   Subjects with normal liver function also need to meet all the following conditions:
3. When screening, the following demographic matching criteria must be met:

   1. Match the weight with the liver function impairment group, with a mean of ± 10 kg;
   2. Age matched with the liver function impairment group, with a mean of ± 10 years;
   3. Gender matching was performed with the liver function impairment group, with a mean of ± 1 case;

   Subjects with liver function impairment also need to meet all the following conditions:
4. Patients with chronic liver injury caused by primary liver diseases (such as hepatitis B, hepatitis C, autoimmune hepatitis, alcoholic liver disease, etc.) and stable liver function (without any liver disease related medical records within 14 days before taking the study drug, except for regular follow-up and medication) with liver dysfunction classified as A or B by Child-Pugh ;
5. Clinically diagnosed as liver cirrhosis;
6. Those who have a stable medication plan for the treatment of liver function damage, complications, and other accompanying diseases for at least 14 days before taking the study drug, and the medication does not need to be adjusted (including medication type, dosage, or frequency); Or those who have not taken medication;
7. Estimated Glomerular filtration rate (eGFR, calculated using the CKD-EPI formula) ≥ 60 mL/min/1.73m2;

Exclusion Criteria:

1. The electrocardiogram shows a QTc interval (QTcF) of>450 msec for males and>470 msec for females (corrected according to Fridericia's standard);
2. Screening for individuals with severe infections, trauma, gastrointestinal surgery, or other major surgical procedures within the first 4 weeks;
3. Those who have received the vaccine within 14 days before screening or plan to receive the vaccine during the study period;
4. Those who donate blood or have a blood loss of ≥ 400 mL within the first 3 months of screening, or intend to donate blood during or within 1 month after the trial;
5. Screening for potent inhibitors or inducers of Pg-P or BCRP that have been used within the previous month (see Attachment 4);
6. Those who have taken a special diet (including dragon fruit, mango, grapefruit, and/or xanthine diet, chocolate) and/or consumed excessive amounts of tea, coffee, grapefruit/grapefruit juice, and/or caffeinated beverages (an average of 8 or more cups per day, 200 mL per cup) within 2 weeks before administration;
7. Screening for alcoholics within the first three months, i.e. those who consume more than 14 units of alcohol per week (1 unit=360 mL of beer, or 45 mL of 40% alcohol or 150 mL of wine) or those who are positive for alcohol screening;
8. Individuals who smoke an average of 10 or more cigarettes per day within the first 3 months of screening;

   Subjects with normal liver function who meet any of the following exclusion criteria need to be excluded:
9. History of liver injury;
10. Individuals who have previously or currently suffered from any clinical serious diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry, and metabolic abnormalities, or any other diseases that may interfere with the test results;
11. Abnormalities in physical examination, vital signs, laboratory examination, 12 lead electrocardiogram, abdominal ultrasound, and other examinations have been determined by the researcher to have clinical significance;
12. Those who are positive in any index screening of hepatitis B surface antigen, hepatitis C antibody or hepatitis C core antigen, HIV antigen/antibody or syphilis antibody;
13. Have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or supplements within 14 days prior to the administration of the study drug;

    Subjects with liver function impairment who meet any of the following exclusion criteria need to be excluded:
14. The subject has any of the following conditions: drug-induced liver injury; History of liver transplantation; And researchers believe that liver cirrhosis
15. During screening, the laboratory test results meet any of the following criteria: (a) alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>5 × ULN; (b) Absolute value of neutrophils (NE #)<1 × 109/L; (c) Hemoglobin (HGB)<80 g/L; (d) Alpha fetoprotein (AFP)>100 ng/mL;
16. Except for the primary liver disease itself, those who have previously or currently suffered from other serious organ system diseases, including but not limited to gastrointestinal, respiratory, renal, neurological, hematological, endocrine, tumor, immune, mental, or cardiovascular diseases or clinical laboratory examination abnormalities, which have clinical significance, and are determined by the research doctor to be unsuitable for participating in this trial;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
The Cmax of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  maximum observed plasma concentration
The AUC0-t of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  area under the curve from time zero to the last measurable concentration
The AUC0-inf of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  area under curve from time zero to infinity
Tmax of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  Time to maximum observed concentration of the main metabolite 116-N1 of JT001;
t1/2 of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  Terminal phase half-life of the main metabolite 116-N1 of JT001;
CL/F of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  The clearance of the main metabolite 116-N1 of JT001;
Vz/F of the main metabolite 116-N1 of JT001; | From time zero up to 72 hours post-dose following oral administration of JT001
  The apparent volume of distribution of the main metabolite 116-N1 of JT001;
The severity of SAE | From Day 1(first dose) to Day7
  The severity of SAE
The Number of participants with SAE | From Day 1(first dose) to Day7
  The Number of participants with SAE
The severity ofclinical symptoms abnormalities(e.g.,Dizziness, headache, nausea, abdominal pain, fatigue, drowsiness） | From Day 1(first dose) to Day7
  The severity ofclinical symptoms abnormalities(e.g.,Dizziness, headache, nausea, abdominal pain, fatigue, drowsiness）
The Number of participantswith abnormal clinical symptoms(e.g.,Dizziness, headache, nausea, abdominal pain, fatigue, drowsiness） | From Day 1(first dose) to Day7
  The Number of participantswith abnormal clinical symptoms(e.g.,Dizziness, headache, nausea, abdominal pain, fatigue, drowsiness）
The severity of vital signs abnormalities | From Day 1(first dose) to Day7
  The severity of Pulse abnormalities
The Number of participantswith abnormal vital signs | From Day 1(first dose) to Day7
  The Number of participantswith abnormal Pulse
The severity of vital signs abnormalities | From Day 1(first dose) to Day7
  The severity of blood pressure abnormalities
The Number of participantswith abnormal vital signs | From Day 1(first dose) to Day7
  The Number of participantswith abnormal blood pressure
The severity of vital signs abnormalities | From Day 1(first dose) to Day7
  The severity of respiration abnormalities
The Number of participantswith abnormal vital signs | From Day 1(first dose) to Day7
  The Number of participantswith abnormal respiration
The severity of vital signs abnormalities | From Day 1(first dose) to Day7
  The severity of body temperature abnormalities
The Number of participantswith abnormal vital signs | From Day 1(first dose) to Day7
  The Number of participantswith abnormal body temperature
The severity of abnormal physical examinations findings | From Day 1(first dose) to Day7
  The severity of abnormal physical examinations findings
The Number of participantswith abnormal physical examinations findings | From Day 1(first dose) to Day7
  The Number of participantswith abnormal physical examinations findings
The severity of abnormal laboratory tests results | From Day 1(first dose) to Day7
  The severity of abnormal laboratory tests results
The Number of participantswith abnormal laboratory tests results | From Day 1(first dose) to Day7
  The Number of participantswith abnormal laboratory tests results
The severity of electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The severity of Heart rate abnormalities
The Number of participants with electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The Number of participants with Heart rate abnormalities
The severity of electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The severity of PR interval abnormalities
The Number of participants with electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The Number of participants with PR interval abnormalities
The severity of electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The severity of QRS interval abnormalities
The Number of participants with electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The Number of participants with QRS interval abnormalities
The severity of electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The severity of QT interval abnormalities
The Number of participants with electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The Number of participants with QT interval abnormalities
The severity of electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The severity of QTcF abnormalities
The Number of participants with electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The Number of participants with QTcF abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Huiyu Lan, Project Director, Study Director — Shanghai Vinnerna Biosciences Co., Ltd.
Locations (1):
- The First Hospital of Jilin University Ethics Committee, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided